CLINICAL TRIAL: NCT01135914
Title: A Canadian 12-month, Prospective, Randomized, Open-label, Multicenter, Laser-controlled Phase IIIb Study Assessing the Efficacy, Safety and Cost-efficacy of Ranibizumab as Combination and Monotherapy in Patients With Visual Impairment Due to Diabetic Macular Edema.
Brief Title: Safety, Efficacy and Cost-efficacy of Ranibizumab (Monotherapy or Combination With Laser) in the Treatment of Diabetic Macular Edema (DME)
Acronym: RESPOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DCA05
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Macular Edema
Keywords: DME; visual impairment; diabetes; macular edema; diabetic macular edema; ranibizumab; laser; photocoagulation; retinopathy; retina
MeSH Terms: conditions — Vision Disorders; Diabetes Mellitus; Macular Edema; Retinal Diseases | interventions — Ranibizumab; Lasers

ARMS (3):
- Combination Therapy (Experimental): Participants received ranibizumab intravitreal injection and laser photocoagulation treatments
  Interventions: Drug: ranibizumab; Procedure: Laser
- Ranibizumab Monotherapy (Experimental): Participants received ranibizumab intravitreal injection therapy only
  Interventions: Drug: ranibizumab
- Laser Monotherapy (Active Comparator): Participants received Laser photocoagulation therapy only
  Interventions: Procedure: Laser

INTERVENTIONS:
Drug: ranibizumab — Ranibizumab 0.5 mg fixed loading dose via intravitreal injection, given once per month for 3 consecutive months (Day 1, Month 1 and Month 2). This treatment could be reapllied, depending on symptoms.
  Arms: Combination Therapy; Ranibizumab Monotherapy
Procedure: Laser — Laser photocoagulation treatment was administered on Day 1. Subsequent laser treatments could be administered if needed, in accordance with Early Treatment Diabetic Retinopathy Study (ETDRS) guidelines.
  Arms: Combination Therapy; Laser Monotherapy

SUMMARY:
To evaluate, specifically within the Canadian medical environment, the efficacy, safety and cost-efficacy of ranibizumab administered either as combination therapy (ranibizumab plus laser photocoagulation), or as monotherapy in comparison with the current standard of care (laser photocoagulation monotherapy), in patients with visual impairment due to DME.

ELIGIBILITY:
Inclusion Criteria:

* Stable Type 1 or Type 2 diabetes mellitus
* Visual impairment due to focal or diffuse DME in at least one eye

Exclusion Criteria:

* Active conditions in the study eye that could prevent the improvement of visual acuity on study treatment
* Active eye infection or inflammation
* History of stroke, renal failure or uncontrolled hypertension

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Canada (20):
  - Calgary Retina Consultants, Calgary, Alberta
  - UBC - Eye Care Center, Vancouver, British Columbia
  - Retina Consultants of Victoria, Victoria, British Columbia
  - Memorial University Health Sciences Centre / Bense Eye Centre, St. John's, Newfoundland and Labrador
  - Victoria General Hospital, Department of Ophthalmology, Halifax, Nova Scotia
  - Ivey Eye Institute, London, Ontario
  - Canadian Centre for Advanced Eye Therapeutics, Mississauga, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - St-Michael's Hospital - Dept of Ophthalmology, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Clinique ChirurgiVision, Drummondville, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital Notre Dame (CHUM), Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Centre Oculaire de Québec, Québec, Quebec
  - Dr.Michel Giunta Clinique Médicale, Sherbrooke, Quebec
  - Saskatoon City Hospital / Spadina Clinic, Saskatoon, Saskatchewan
  - Institut de l'oeil des Laurentides, Québec
  - Memorial University Health Sciences Centre / Newfoundland Drive Medical Clinic, St. John's

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 239 patients were enrolled in the study. An additional 2 patients were enrolled but were removed from the database because consent was not signed in accordance with GCP principles."
Pre-assignment Details: 3 treatment arms: Group C - laser photocoagulation per ETDRS guidelines, Group B - ranibizumab intravitreal injections (3 monthly injections during loading phase, and subsequent treatments per protocol-defined criteria), or Group A - combination therapy, where decisions to treat with laser were independent of decisions to treat with ranibizumab.
Groups:
- Combination Therapy: Participants received both a ranibizumab intravitreal injection and laser photocoagulation treatments.
Period: Overall Study
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Started | 78 | 80 | 81
Intent to Treat (ITT) Population | 73 | 75 | 72
Safety Population | 73 | 75 | 74
Completed | 74 | 75 | 59
Not Completed | 4 | 5 | 22
Not completed — Withdrawal by Subject | 1 | 3 | 6
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 3
Not completed — Lack of Efficacy | 2 | 1 | 10
Not completed — Adverse Event | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) population was defined as all patients receiving at least one dose of either study treatment for monotherapy treatment arms, or one of the two study treatments for the combination therapy arm, and having at least 1 post-baseline assessment. Patients from a center were excluded from ITT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy | Total
Number analyzed (Participants) | 73 | 75 | 72 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.21) | 61.5 (9.86) | 62.8 (9.44) | 61.7 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 29 | 88
  Male | 47 | 42 | 43 | 132

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity- (BCVA) at Month 12
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of BCVA (EDTRS) is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement.
Time Frame: Baseline and 12 months
Population: ITT defined as all patients receiving at least one dose of either study treatment for monotherapy treatment arms, or one of the two study treatments for the combination therapy arm, and having at least 1 post-baseline assessment. Patients from one study site were excluded from ITT. patients with both baseline and 12 month data were included.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 70 | 71 | 62
Letters | 8.2 (9.20) | 8.9 (7.78) | 0.3 (12.47)

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Months 3,6 and 9
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of BCVA (EDTRS)is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement.
Time Frame: Baseline, 3, 6 and 9 months
Population: The ITT population was defined as all patients receiving at least one dose of either study treatment for monotherapy treatment arms, or one of the two study treatments for the combination therapy arm, and having at least 1 post-baseline assessment. Patients from one site were excluded from ITT.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 73 | 75 | 72
Letters
  Month 3 (n=71, 75, 69) | 3.7 (10.71) | 5.3 (7.58) | 1.4 (6.55)
  Month 6 (n= 70, 72, 65) | 5.6 (8.45) | 7.1 (7.74) | 0.9 (7.23)
  Month 9 (n=69, 71, 59) | 7.1 (7.92) | 6.9 (12.45) | -0.2 (10.71)

3. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Months 3,6,9 and 12
Description: OCT is a diagnostic imaging technique using low-coherence interferometry to produce cross-sectional tomograms of the posterior segment eye structures. OCT was performed prior to study treatment to assess CRT, presence of fluid in the macula (intra-retinal cyst or fluid) and evaluation of image to monitor disease progression/treatment effect and to determine the need to stop/re-initiate ranibizumab treatment
Time Frame: Baseline, 3, 6, 9 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 73 | 75 | 72
um
  Baseline | 422.1 (142.26) | 448.5 (136.64) | 458.0 (133.07)
  Month 3 (n=71,75, 69) | -105.7 (127.74) | -108.9 (113.38) | -32.5 (114.15)
  Month 6 (n= 70,72,65) | -114.2 (110.88) | -129.3 (116.50) | -64.4 (110.77)
  Month 9 (69,70,58) | -138.1 (125.86) | -135.9 (140.90) | -85.8 (128.00)
  Month 12 (70,71,61) | -152.2 (139.27) | -143.5 (143.95) | -107.1 (143.86)

4. Secondary Outcome: Percentage of Patients Achieving a Gain of 15-letters or More (3-lines) in BCVA From Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of BCVA (EDTRS) is 0 to 100 letters. A higher percent of patients achieving a gain of ≥15 letters BCVA indicates a better response.
Time Frame: Baseline, 3, 6, 9 and 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 73 | 75 | 72
Percentage of Patients
  Month 3 (n=71,75,69) | 8.5 | 9.3 | 2.9
  Month 6 (n=70,72,65) | 11.4 | 13.9 | 1.5
  Month 9 (69,71,59) | 13.0 | 21.1 | 0
  Month 12 (70,71,62) | 24.3 | 21.1 | 6.5

5. Secondary Outcome: Percentage of Patients Achieving Gain of Letters From Baseline in BCVA
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of BCVA (EDTRS) is 0 to 100 letters. A gain of 5,10,15 or more BCVA letters from baseline indicates improvement.
Time Frame: 12 months
Population: ITT defined as all patients receiving at least one dose of either study treatment for monotherapy treatment arms, or one of the two study treatments for the combination therapy arm, and having at least 1 post-baseline assessment. Patients from one study site were excluded from ITT. Patients with 12 month data were included
Measure: Number; unit: Percentage of Patients
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 70 | 71 | 62
Percentage of Patients
  5 letter gain | 61.4 | 70.4 | 40.3
  10 letter gain | 34.3 | 52.1 | 16.1
  15 letter gain | 24.3 | 21.1 | 6.5

6. Secondary Outcome: National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25) Composite Score at Month 12
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) was used to measure the influence of visual disability and visual symptoms on general health domains. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. For each question, the patient was asked to rate their condition on a scale of 1-5 or 1-6, where a low number reflects a better outcome. A composite score for a patient is calculated by aggregating and averaging the scores from the 11 sub-scales (excluding general health sub-scale), and an algorithm is apply to give equal weight to each sub-scale. Sub-scales and composite scores are calculated by converting the response from questionnaires into a 0-100 scale, with 0 as the worst possible outcome and 100 as the best. Missing data was not imputed
Time Frame: 12 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 70 | 71 | 62
Units on a Scale | 85.21 (12.77) | 84.29 (11.78) | 78.20 (17.27)

7. Secondary Outcome: EuroQoL (EQ-5D) Utility Score at Month 12
Description: The Euro Quality of Life Questionnaire (EQ-5D) standardized instrument was utilized to measure health outcomes related to 5 dimensions, namely: mobility, self-care, usual activities, pain-discomfort, and anxiety/depression. The possible range for each dimension was 1 to 3, where 1="no problems", 2="some problems" and 3="extreme problems". Missing values were not imputed. Using the scoring algorithm derived from the Canadian value sets (Bansback et al., 2012), a utility score for a patient was calculated based on the EQ-5D responses for a given time-point at which the questionnaire was presented to the patient. This mean EQ-5D utility score ranged between 0 (worst health) to 1 (perfect health).
Time Frame: 12 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 68 | 71 | 60
Units on a scale | 0.88 (0.15) | 0.88 (0.17) | 0.87 (0.17)

8. Secondary Outcome: Time Trade-Off Questionnaire - 25 (TTO) Composite Score at Month 12
Description: (TTO) questionnaire was used to help determine the patients' health utility. Reported health utility represents the patients' quality of life at the current health state, and is a cardinal value that ranges from 0 (worst possible health or death) to 1 (best possible health). In this questionnaire, patients were first asked to estimate their remaining life expectancy. Second, the patients were presented with a hypothetical situation where a technology existed that could permanently return their vision to normal. This technology would always work, but would decrease their length of survival. Patients were then asked how much of their remaining life expectancy, if any, they would be willing to trade in return for use of the technology and thus for normal vision. The principle of this measure is that if patients were content with their current vision status (i.e., have a utility value of 1.0), they would not want to trade any of their remaining life years to improve their vision.
Time Frame: 12 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Number analyzed (Participants) | 69 | 68 | 60
Units on a scale | 0.83 (0.28) | 0.78 (0.23) | 0.80 (0.24)

ADVERSE EVENTS:
Description: The Safety population was defined as all patients who received at least 1 administration of ranibizumab/laser treatment for monotherapy, or at least one of the two treatments for combination therapy, excluding patients from one site
Arm/Group | Combination Therapy | Ranibizumab Monotherapy | Laser Monotherapy
Serious Adverse Events (participants affected / at risk) | 9/73 | 10/75 | 5/74
Other Adverse Events (participants affected / at risk) | 26/73 | 26/75 | 17/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=73) | Ranibizumab Monotherapy (N=75) | Laser Monotherapy (N=74)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 0 | 0 | 2
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=73) | Ranibizumab Monotherapy (N=75) | Laser Monotherapy (N=74)
Cataract (Fellow eye) (Eye disorders) | 0 | 5 | 3
Cataract (Study eye) (Eye disorders) | 0 | 5 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 9 | 6 | 1
Eye irritation (Study eye) (Eye disorders) | 4 | 0 | 0
Vision blurred (Study eye) (Eye disorders) | 4 | 0 | 0
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 4 | 2 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 0 | 4
Nasopharyngitis (Infections and infestations) | 5 | 5 | 4
Intraocular pressure increased (Fellow eye) (Investigations) | 4 | 4 | 3
Intraocular pressure increased (Study eye) (Investigations) | 8 | 10 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Headache (Nervous system disorders) | 1 | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 5 | 1 | 0
Hypertension (Vascular disorders) | 2 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e. data from all sites) in the clinical trial or dislcosure of trial results in their entirety.